CLINICAL TRIAL: NCT03309722
Title: Molecular Pathology of Colorectal Cancer: Investigating the Role of Novel Molecular Profiles, microRNA's, and Their Targets in Colorectal Cancer
Brief Title: Molecular Pathology of Colorectal Cancer: Investigating the Role of Novel Molecular Profiles, microRNA's, and Their Targets in Colorectal Cancer Progression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: UKCRNID6067
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early stage
  Interventions: Other: biomarker study
- advanced
  Interventions: Other: biomarker study

INTERVENTIONS:
Other: biomarker study

SUMMARY:
Molecular pathology of Colorectal Cancer: Investigating the role of novel molecular profiles, microRNA's and their targets in Colorectal Cancer progression

DETAILED DESCRIPTION:
Single centre observational cohort study Prospectively recruited patients biomarker evaluation and identification of novel biomarkers

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer

Exclusion Criteria:

* hereditary CRC; tumours with extensive necrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with colorectal cancer that consent to study and fit inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-10-10 (Actual); Primary Completion 2020-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
disease free survival | 5 years
local recurrence | 5 years
distant recurrence | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Hanley CJ, Noble F, Ward M, Bullock M, Drifka C, Mellone M, Manousopoulou A, Johnston HE, Hayden A, Thirdborough S, Liu Y, Smith DM, Mellows T, Kao WJ, Garbis SD, Mirnezami A, Underwood TJ, Eliceiri KW, Thomas GJ. A subset of myofibroblastic cancer-associated fibroblasts regulate collagen fiber elongation, which is prognostic in multiple cancers. Oncotarget. 2016 Feb 2;7(5):6159-74. doi: 10.18632/oncotarget.6740. PMID 26716418
- [Background] Cellura D, Pickard K, Quaratino S, Parker H, Strefford JC, Thomas GJ, Mitter R, Mirnezami AH, Peake NJ. miR-19-Mediated Inhibition of Transglutaminase-2 Leads to Enhanced Invasion and Metastasis in Colorectal Cancer. Mol Cancer Res. 2015 Jul;13(7):1095-1105. doi: 10.1158/1541-7786.MCR-14-0466. Epub 2015 May 1. PMID 25934693
- [Background] Ling H, Pickard K, Ivan C, Isella C, Ikuo M, Mitter R, Spizzo R, Bullock M, Braicu C, Pileczki V, Vincent K, Pichler M, Stiegelbauer V, Hoefler G, Almeida MI, Hsiao A, Zhang X, Primrose J, Packham G, Liu K, Bojja K, Gafa R, Xiao L, Rossi S, Song JH, Vannini I, Fanini F, Kopetz S, Zweidler-McKay P, Wang X, Ionescu C, Irimie A, Fabbri M, Lanza G, Hamilton SR, Berindan-Neagoe I, Medico E, Mirnezami A, Calin GA, Nicoloso MS. The clinical and biological significance of MIR-224 expression in colorectal cancer metastasis. Gut. 2016 Jun;65(6):977-989. doi: 10.1136/gutjnl-2015-309372. Epub 2015 Mar 24. PMID 25804630
- [Background] Bullock MD, Pickard K, Mitter R, Sayan AE, Primrose JN, Ivan C, Calin GA, Thomas GJ, Packham GK, Mirnezami AH. Stratifying risk of recurrence in stage II colorectal cancer using deregulated stromal and epithelial microRNAs. Oncotarget. 2015 Mar 30;6(9):7262-79. doi: 10.18632/oncotarget.3225. PMID 25788261
- [Background] Bullock MD, Mellone M, Pickard KM, Sayan AE, Mitter R, Primrose JN, Packham GK, Thomas G, Mirnezami AH. Molecular profiling of the invasive tumor microenvironment in a 3-dimensional model of colorectal cancer cells and ex vivo fibroblasts. J Vis Exp. 2014 Apr 29;(86):51475. doi: 10.3791/51475. PMID 24836208
- [Background] Zhang L, Pickard K, Jenei V, Bullock MD, Bruce A, Mitter R, Kelly G, Paraskeva C, Strefford J, Primrose J, Thomas GJ, Packham G, Mirnezami AH. miR-153 supports colorectal cancer progression via pleiotropic effects that enhance invasion and chemotherapeutic resistance. Cancer Res. 2013 Nov 1;73(21):6435-47. doi: 10.1158/0008-5472.CAN-12-3308. Epub 2013 Aug 15. PMID 23950211